CLINICAL TRIAL: NCT01214980
Title: A Prospective, Randomized, Controlled Pilot Study of the MIST Therapy System for the Treatment of Split Thickness Donor Sites
Brief Title: Split Thickness Donor Site Healing With MIST Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celleration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-86003
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Burns; Trauma; Venous Ulcers
Keywords: Low-frequency ultrasound; Wound healing; Split thickness wound healing; Skin graft donor site healing
MeSH Terms: conditions — Burns; Wounds and Injuries; Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MIST Therapy in conjunction with SOC (Experimental): Low-frequency, non-contact ultrasound administered in conjunction with standard of care treatment
  Interventions: Device: MIST Therapy
- Control arm (Active Comparator): Standard of care treatment
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: MIST Therapy — Low-frequency, non-contact ultrasound therapy provided in conjunction with standard of care treatment on a daily basis for 5 days.
  Other Names: MIST; MIST Treatment
  Arms: MIST Therapy in conjunction with SOC
Other: Standard of care — Standard of care provided per site-specific protocol
  Other Names: Standard wound care
  Arms: Control arm

SUMMARY:
Subjects requiring skin grafting due to burns, trauma, or chronic venous ulcers with split thickness donor sites expected to be between 20 and 200 square cm will be consecutively screened for study eligibility. This study is a prospective, randomized, controlled trial evaluating effect of MIST Therapy on the healing of split thickness skin graft donor sites compared to standard care. Subjects meeting all eligibility criteria and providing appropriate written informed consent will be enrolled for study participation.

DETAILED DESCRIPTION:
Enrolled subjects will be randomized to receive one of two treatment courses: a) MIST Therapy in conjunction with standard of care (SOC) (treatment group); or b)SOC alone (control group).

On post-op day 1, subjects will undergo a baseline evaluation prior to initiating assigned study treatment, including: wound measurement, wound bed evaluation, description of periwound skin, measurement of type and quantity of exudation, wound clinical symptoms (pain, burning, itching), and digital photography. Subject will then receive assigned study treatment.

SOC includes, but is not limited to, fluid resuscitation, pain medications, systemic antibiotics, control of bleeding, and standard dressings as appropriate for the moisture balance of the wound. SOC also includes providing a hydrocolloid border around the wound with a transparent film dressing over the donor site. No advanced or impregnated dressings are allowed during the study. No topical antibiotics or antibiotic dressings, topical antiseptics (silver, iodine, etc.,) or antimicrobials are allowed.

The transparent film will be removed each day and wound fluid will be collected for analysis. After wound fluid collection, subjects will receive their assigned study treatment. Subjects randomized to receive MIST Therapy will be treated daily for 5 consecutive days. Following administration of the assigned study treatment, subjects will have replacement of the transparent film. The hydrocolloid will remain in place on the border of intact skin.

Evaluations performed will include a wound assessment, digital photography, wound pain assessment and an adverse event assessment. Following the initial 5 day treatment, the study wounds will be dressed per SOC with dressing changes as needed.

Subjects will undergo a weekly wound assessment through 6 weeks from the date of study enrollment. A weekly wound assessment will include the assessment of maintained wound closure, digital photography, and an adverse event assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject of any race and at least 18 years old
* Subject requires skin grafting
* Subject's wound must be between 20 cm2 and 200 cm2
* Subject's wound presents with no clinical signs of acute infection
* Subject has ahd no prior MIST Therapy to the enrolled wound
* Subject or subject's legally authorized representative understands the nature of the procedure(s) and provides written informed consent prior to study enrollment
* Subject is willing and able to comply with all specified care and visit requirements
* Women of childbearing potential must not be pregnant or lactating, and must be using adequate and accepted contraceptive methods
* Subject has a reasonable expectation of completing the study

Exclusion Criteria:

* Subject's condition requires the use of topical antibiotics at the time of study enrollment
* Subject's wound would require ultrasound near an electronic implant or prosthesis, e.g., near or over the heart, or over the thoracic area if the subject is using a cardiac pacemaker
* Subject is known to be suffering from a disorder or other situation that the subject or investigator feels would interfere with compliance or other study requirements
* Subject is currently enrolled or has been enrolled in the last 30 days in another investigational device or drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Gould, M.D.,Ph.D, Principal Investigator — James A. Haley Veterans Hospital; David Smith, MD, Principal Investigator — University South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

REFERENCES:
- [Derived] Sinha S, Gabriel VA, Arora RK, Shin W, Scott J, Bharadia SK, Verly M, Rahmani WM, Nickerson DA, Fraulin FO, Chatterjee P, Ahuja RB, Biernaskie JA. Interventions for postburn pruritus. Cochrane Database Syst Rev. 2024 Jun 5;6(6):CD013468. doi: 10.1002/14651858.CD013468.pub2. PMID 38837237
- [Derived] Prather JL, Tummel EK, Patel AB, Smith DJ, Gould LJ. Prospective Randomized Controlled Trial Comparing the Effects of Noncontact Low-Frequency Ultrasound with Standard Care in Healing Split-Thickness Donor Sites. J Am Coll Surg. 2015 Aug;221(2):309-18. doi: 10.1016/j.jamcollsurg.2015.02.031. Epub 2015 Mar 14. PMID 25868409

RESULTS

PARTICIPANT FLOW:
Groups:
- MIST Therapy in Conjunction With Standard Care: Low-frequency, non-contact ultrasound administered in conjunction with standard of care treatment
  MIST Therapy: Low-frequency, non-contact ultrasound therapy provided in conjunction with standard of care treatment (Wound cleansing followed by application of a hydrocolloid border and a transparent dressing for a moist wound environment that allows for dressing removal without trauma) on a daily basis for 5 days.
- Control Arm: Standard of care treatment
  Standard of care: Standard of care provided per site-specific protocol Wound cleansing followed by application of a hydrocolloid border and a transparent dressing for a moist wound environment that allows for dressing removal without trauma
Period: Overall Study
Arm/Group | MIST Therapy in Conjunction With Standard Care | Control Arm
Started | 16 | 16
Completed | 13 | 14
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | MIST Therapy in Conjunction With Standard Care | Control Arm | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Median (Full Range); unit: years] | 32 [20 to 91] | 54 [25 to 82] | 49 [20 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 11 | 11 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 12 | 12 | 24
  Hispanic/Latino | 0 | 1 | 1
  African American | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
BMI [Median (Full Range); unit: kilograms per meter squared] | 24.7 [16.8 to 41.1] | 25.0 [20.3 to 34.0] | 24.7 [16.8 to 41.4]
Number of donor sites [Median (Full Range); unit: number of sites] | 2 [1 to 4] | 1.5 [1 to 5] | 2 [1 to 5]
Baseline donor site size [Median (Full Range); unit: centimeters squared] | 139.5 [36.0 to 200.0] | 136.0 [36.0 to 216.0] | 136.0 [36.0 to 216.0]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Wound Healing
Description: The primary endpoint is an average of the group for each participant's donor site wound closure time, defined as days to absence of drainage from the date of the initial donor site harvest procedure.
Time Frame: Days to absence of drainage from the initial donor site harvest procedure
Population: randomized participants that had a minimum of 4 out of 5 treatments
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MIST Therapy in Conjunction With Standard Care | Control Arm
Number analyzed (Participants) | 13 | 14
Days | 12.1 (6.0) | 21.3 (14.7)

2. Secondary Outcome: Time to Full Epithelialization
Description: Time to full epithelialization in days from the date of initial donor site harvest procedure per the blinded adjudication of the donor site image.
Time Frame: Days to full epithelialization
Population: randomized subjects that had a minimum of 4 out of 5 study treatments
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MIST Therapy in Conjunction With Standard Care | Control Arm
Number analyzed (Participants) | 13 | 14
days | 18.2 (8.8) | 27.5 (12.2)

3. Secondary Outcome: Numeric Pain Score
Description: Average donor site pain score for each treatment group, numeric scale of 0 (no pain) to 10 (worst possible pain), at five weeks post skin graft procedure
Time Frame: 5 weeks
Population: randomized subjects that had a minimum of 4 out of 5 study treatments and with a numeric pain score reported
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MIST Therapy in Conjunction With Standard Care | Control Arm
Number analyzed (Participants) | 10 | 10
units on a scale | 0 (.964) | 1.8 (.964)

4. Secondary Outcome: Numeric Itching Score
Description: Average donor site itching score for treatment group, numeric scale 0 (no itch) to 10 (worst possible itch), at 5 weeks post skin graft procedure
Time Frame: 5 weeks
Population: Randomized subjects with a minimum of 4 out of 5 study treatments and itching score reported
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MIST Therapy in Conjunction With Standard Care | Control Arm
Number analyzed (Participants) | 10 | 9
units on a scale | 0.7 (1.3) | 4.1 (1.3)

5. Secondary Outcome: Donor Site Recidivism Rate
Description: Number of donor sites that healed and then reopened during the study.
Time Frame: 6 weeks
Population: Randomized subjects that had a minimum of 4 out of 5 study treatments and fully epithelialized during the study.
Measure: Number; unit: participants that healed and reopened
Arm/Group | MIST Therapy in Conjunction With Standard Care | Control Arm
Number analyzed (Participants) | 13 | 11
participants that healed and reopened | 1 | 5

ADVERSE EVENTS:
Time Frame: 6 weeks post skin graft procedure
Description: Device related events and infections
Arm/Group | MIST Therapy in Conjunction With Standard Care | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 4/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIST Therapy in Conjunction With Standard Care (N=16) | Control Arm (N=16)
Infection (Infections and infestations) | 1 (1) | 4 (4) — Infection of the donor site wound
Discomfort (General disorders) | 3 (3) | 0 (0) — Discomfort with repositioning / treatment

LIMITATIONS AND CAVEATS:
Participants were not blinded to study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No